CLINICAL TRIAL: NCT05515822
Title: Use of Oxycodone in Multimodel Perioperative Analgesia of Bariatric Surgery and Its Effect on Inflammatory Factors
Brief Title: Use of Oxycodone in Bariatric Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qiang Fu (Other)
Responsible Party: Sponsor-Investigator, Qiang Fu, Chief Physician of Anesthesiology Department, The Third People's Hospital of Chengdu
Organization: The Third People's Hospital of Chengdu (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ezmr2022-018
Record Dates: First submitted 2022-08-21; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Pain, Postoperative
Keywords: Oxycodone; Acute Postoperative Pain; clinical randomized trial
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxycodone; dezocine; Esketamine

STUDY DESIGN:
Intervention Model Description: Control group: Dezocine +Patient-controlled intravenous analgesia (Dezocine) ; Intervention group A: Oxycodone +Patient-controlled intravenous analgesia (Oxycodone); Intervention group B: Esketamine + Oxycodone +Patient-controlled intravenous analgesia (Oxycodone) .
Who Masked: Participant, Care Provider
Masking Description: Random numbers and groups are packed in opaque envelopes. The experimenter will open an envelope according to the random number on the envelope cover in the order from small to large according to the time of inclusion of the subject, and then obtain the random grouping of the subject (1:1:1). The random number is generated by computer, sealed into an envelope, unsealed and dispensed by professionals who do not participate in test operations. Participants and postoperative visitors did not know the grouping information. In emergency situations (e.g. allergies) or after data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dezocine group (Active Comparator): Dezocine (1ml: 5mg) was administered 30 minutes before the end of surgery (0.15mg/kg i.v.) and during patient controlled intravenous analgesia (Dezocine 30mg+ Tropisetron 10mg+Saline, total 200ml)
  Interventions: Drug: Dezocine
- Oxycodone group (Experimental): Oxycodone (1ml: 10mg) was administered 30 minutes before the end of surgery (0.15mg/kg i.v.) and during patient controlled intravenous analgesia (Oxycodone 30mg+ Tropisetron 10mg+Saline, total 200ml)
  Interventions: Drug: Oxycodone Hydrochloride
- Esketamine+Oxycodone group (Experimental): Esketamine (2ml: 50mg) was administered 5 minutes before incision (0.15mg/kg i.v.), while Oxycodone was administered 30 minutes before the end of surgery (0.15mg/kg i.v.) and during patient controlled intravenous analgesia (Oxycodone 30mg+ Tropisetron 10mg+Saline, total 200ml)
  Interventions: Drug: Esketamine and Oxycodone

INTERVENTIONS:
Drug: Oxycodone Hydrochloride — The doses were calculated according to the ideal body weight. Oxycodone was administered within 30min before the end of surgery. The parameters of patient controlled intravenous analgesia (PCIA) pump were set as continuous volume: 0ml, PCA: 6ml, lock time: 5min, extreme limit: 30ml, and connect with peripheral venous access at the beginning of skin suture.
  Other Names: Oxycodone group; Experimental
  Arms: Oxycodone group
Drug: Dezocine — Dezocine was administered within 30min before the end of surgery. The parameters of patient controlled intravenous analgesia (PCIA) pump were set as continuous volume: 0ml, PCA: 6ml, lock time: 5min, extreme limit: 30ml, and connect with peripheral venous access at the beginning of skin suture.
  Other Names: Dezocine group; Active Comparator
  Arms: Dezocine group
Drug: Esketamine and Oxycodone — Esketamine was administered 5min before skin incision, and Oxycodone was administered within 30min before the end of surgery. The parameters of patient controlled intravenous analgesia (PCIA) pump were set as continuous volume: 0ml, PCA: 6ml, lock time: 5min, extreme limit: 30ml, and connect with peripheral venous access at the beginning of skin suture.
  Other Names: Esketamine+Oxycodone group; Experimental
  Arms: Esketamine+Oxycodone group

SUMMARY:
There is still no effective treatment for surgical pain, especially visceral pain in bariatric surgery. Oxycodone has great application prospect in patients with obesity, but there are few clinical studies and analgesic effect is still unclear, especially in combination with esketamine.

This study was a prospective, single-center, randomized, controlled, double-blind clinical trial to compare the efficacy and safety of intravenous oxycodone and combined use of esketamine for perioperative multimodel analgesia during bariatric surgery, and the effect of esketamine on inflammatory factors.

This study was based on the hypothesis that oxycodone and the combination use with esketamine can effectively reduce the level of postoperative pain and inflammatory factors, and does not increase perioperative adverse reactions in bariatric surgery.

DETAILED DESCRIPTION:
The ideal analgesia for bariatric surgery in obese individuals is one that provides effective analgesia for gastrointestinal trauma and abdominal wall incisions without inhibiting respiratory and gastrointestinal recovery. Although many researches have been done on surgical analgesia, there is still no very effective treatment for pain caused by surgery, especially visceral pain.

Oxycodone is a new type of opioid with pure μ and κ receptor double agonists. κ-receptor agonist has specific analgesic effect on visceral pain. Studies have found that oxycodone has obvious effect on visceral pain after abdominal surgery, and at the same time, oxycodone almost does not affect respiration and gastrointestinal peristalsis, which has great application prospect in obese people. However, opioids (including oxycodone) can cause drug tolerance and hyperalgesia, which may be mediated by NMDA receptor activation in the central nervous system. Esketamine provides exact analgesic effect by antagonizing NMDA receptors, with mild respiratory depression and less gastrointestinal and psychiatric adverse reactions. As an analgesic adjuvant, it can reduce the consumption of opioids and increase the analgesic effect when used in combination with other drugs.

Therefore, a prospective, single-center, randomized, controlled, double-blind trial was designed to compare the efficacy and safety of intravenous oxycodone plus esketamine for perioperative multimodal analgesia and the effects on inflammatory cytokines levels during bariatric surgery.

Participants were divided into an intervention group with oxycodone or (and) esketamine, and a control group with dezocine. The main concerns are the effectiveness of postoperative analgesia and the occurrence of adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥30kg/m2;
* Laparoscopic sleeve gastrectomy (LSG) was performed;
* American Society of Anesthesiologists (ASA) Grade I to II, age: 18-50;
* Patient-controlled intravenous analgesia (PCIA) was approved.

Exclusion Criteria:

* Do not agree to sign informed consent or cannot sign for other reasons;
* Oxycodone contraindications;
* Patients with contraindications to esketamine;
* Disocine contraindications;
* Preoperative history of opioid allergy and abuse;
* Have a long history of alcoholism;
* A history of surgery or anesthesia recently;
* Changes in standard anesthesia procedures for any reason.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in postoperative pain | Within 48 hours after surgery.
  The Visual analogue Scale (VAS) was used to evaluate the intensity of postoperative resting state, motor state, and visceral pain within 48 hours after surgery. VAS ranges from 0 to 10, where 0 represents no pain and 10 represents excruciating pain, with higher scores indicating greater pain.
Postoperative opioid consumption | Within 48 hours after surgery.
  The total postoperative opioid consumption was recorded within 48 hours after surgery. Postoperative opioid consumption was evaluated using intravenous morphine equivalent (IVME).

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | Within 48 hours after surgery.
  Postoperative nausea and vomiting (PONV) was evaluated within 48 hours after surgery. 11-point verbal numeric rating scale (VNRS) was used to evaluate nausea (none:0, mild: 1-3, moderate:4-6, severe 7-10). Vomiting was considered a condition of retching symptom or the presence of vomit.
Time to extubation | Intraoperative (From the end of surgery to the removal of the endotracheal tube)
  The total extubation time from the end of surgery to the removal of the endotracheal tube was evaluated after surgery.
Ramsay sedation score | Within 48 hours after surgery.
  Ramsay sedation score was evaluated within 48 hours after surgery. Ramsay sedation score from 1 to 6, with higher scores indicating deeper the sedation.
Finger pulse oxygen saturation (SpO2) | Within 48 hours after surgery.
  Finger pulse oxygen saturation (SpO2) was evaluated within 48 hours after surgery.
Adverse effect | During the hospital stay after surgery, an expected average of three days.
  Perioperative adverse effects such as shivering, blurred vision, headache, dizziness, dry mouth, respiratory depression during postoperative to discharge.
Total amount of anesthetic drugs used | Intraoperative (During the whole bariatric surgery)
  Total amount of anesthetic drugs Propofol, Remifentanil and (or) sevoflurane used was evaluated during the whole surgery.
Total length of stay | During the hospital stay after surgery, an expected average of three days.
  Total length of stay was evaluated from postoperative to discharge.
First time to get out of bed after surgery | During the hospital stay after surgery, an expected average of three days.
  First time to get out of bed after surgery was evaluated after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Fu, Principal Investigator — The Third People's Hospital of Chengdu

IPD SHARING:
Plan to Share IPD: No
The results of the study will be published in the form of a paper, and the information of specific participants will be kept confidential.